CLINICAL TRIAL: NCT02801188
Title: Evaluation Effect of Adding Dexmedetomidine to Bupivacaine for Paravertebral Block in Femoral Fractures
Brief Title: Effect of Dexmedetomidine and Bupivacaine for Paravertebral Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD ∕ 128
Record Dates: First submitted 2016-04-22; First posted 2016-06-15 (Estimated); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Fracture of Proximal Femur
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine group (Placebo Comparator): Paravertebral blockade will be performed using combined mixture of bupivacaine 0.5% and water soluble radio-opaque dye.
  Interventions: Drug: Bupivacaine
- Mixture of bupivacaine and dexmedetomidine group (Active Comparator): Paravertebral blockade will be performed using combined mixture of bupivacaine 0.5%, water soluble radio-opaque dye and 1 ug/kg of dexmedetomidine
  Interventions: Drug: Mixture of bupivacaine and dexmedetomidine

INTERVENTIONS:
Drug: Bupivacaine — Paravertebral blockade will be performed using combined mixture of bupivacaine 0.5% and water soluble radio-opaque dye.
  Arms: Bupivacaine group
Drug: Mixture of bupivacaine and dexmedetomidine — Paravertebral blockade will be performed using combined mixture of bupivacaine 0.5%, water soluble radio-opaque dye, and1 ug/kg of dexmedetomidine
  Arms: Mixture of bupivacaine and dexmedetomidine group

SUMMARY:
Fracture femur is a common that results in severe pain. Many methods of regional and peripheral analgesia have been described to treat such pain. In this study the investigators consider using paravertebral block to treat post-fracture pain. Additionally, they consider adding dexmedetomidine to the used local anesthetic solution to prolong the duration of this block and hence postoperative analgesia.

DETAILED DESCRIPTION:
Fracture femur is a common injury which is associated with excruciating pain . This pain is one of the most important causes of postoperative morbidity and mortality when it is insufficiently treated pain. Pain induces neuroendocrine stress response causing problems like as reduction in vital capacity, pneumonia, tachycardia, hypertension, myocardial ischemia and even infarction. These problems can be prevented by successful management of postoperative pain.

In patients with proximal femoral fracture, the use of paravertebral blockade produces reliable level of analgesia without need for additional nursing skills or monitoring in the postoperative period. Paravertebral blockade by injection local anesthetic solution alongside the vertebral column produces ipsilateral analgesia.

Currently available local anesthetics as bupivacaine may not provide reliable periods of analgesia resulting in block resolution before the period of worst postoperative pain. The use of a large volume of local anesthetic is one of methods to overcome this problem that may lengthen the duration of analgesia but at increased risk of local anesthetic toxicity. Adding adjuvants is another potential alternative.

Dexmedetomidine, a selective α 2 agonist, has been used to prolong the duration of analgesia of nerve blocks. Dexmedetomidine has also been reported to enhance central and peripheral nerve blockade. Alpha adrenoceptors located at the nerve endings have a possible role in the analgesic mechanisms by preventing norepinephrine release. The spinal mechanism is the principle mechanism for the analgesic action of dexmedetomidine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical class I or II

Exclusion Criteria:

* Patient refusal.
* Severe or uncompensated cardiovascular disease.
* Severe or uncompensated renal disease.
* Severe or uncompensated hepatic disease.
* Severe or uncompensated endocrinal disease.
* Pregnancy.
* Postpartum ladies.
* Lactating females.
* Allergy to any of the study medications .
* Coagulation disorders.
* Infection at the site of needle insertion

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Scale for radiological spread of the injectate | for 20 min after performing the blockade
  It will be assessed using the following scale -2; spread for two vertebral levels below the site of injection, -1; spread for one vertebral level below the site of injection, 0; stays at the level of injection, +2; spread for two vertebral levels above the site of injection, +1; spread for one vertebral level above the site of injection

SECONDARY OUTCOMES:
Pain scores | For 48 hours after surgery
  The severity of pain will be assessed using a visual analog scale (VAS)
Duration of postoperative analgesia | for 24 hours after surgery
  The period from completion of the block to time of administration of the first request of rescue analgesic for postoperative pain will be recorded
Postoperative analgesic consumption | for 48 hours after surgery
  Total postoperative analgesic consumption

CONTACTS AND LOCATIONS:
Overall Officials: Reem A El sharkawy, MD, Principal Investigator — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt; Mohamed Y Makharita, MD, Study Director — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt; Nabil Abd-El Raouf, MD, Study Chair — Department of Anaesthesia, Surgical Intensive Care and Pain Medicine, College of Medicine, Mansoura University, Mansoura, Egypt
Locations (1):
- Mansoura university, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided